CLINICAL TRIAL: NCT04294563
Title: Peanut Protein Supplementation to Prevent Muscle Atrophy and Improve Recovery Following Total Knee Arthroplasty
Status: Terminated | Phase: Not Applicable | Type: Interventional
Why Stopped: Accrual targets not met
Sponsor: Auburn University (Other)
Collaborators: Edward Via College of Osteopathic Medicine-Auburn (Unknown); Jack Hughston Memorial Hospital (Unknown)
Responsible Party: Principal Investigator, Andrew Fruge, Assistant Professor and DPD Director, Auburn University
Allocation: Randomized | Model: Parallel | Masking: Triple | Purpose: Supportive Care
Other Study IDs: AU 20-104
Record Dates: First submitted 2020-03-01; First posted 2020-03-04 (Actual); Last update posted 2023-04-21 (Actual); Status verified 2023-04

CONDITIONS: Surgery
Keywords: total knee arthroplasty; physical rehabilitation; protein supplementation; muscular atrophy; inflammatory cytokines
MeSH Terms: conditions — Muscular Atrophy | interventions — Physical Therapists

STUDY DESIGN:
Who Masked: Care Provider, Investigator, Outcomes Assessor
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- Immediate Intervention Group (Experimental): Participants will complete baseline measures and begin daily supplementation of peanut protein powder (72g/day) 7 days prior to total knee arthroplasty until 6 weeks after surgery.
  Interventions: Dietary Supplement: Peanut Protein Powder; Other: Standard Care by Surgeon and Physical Therapist
- Wait-llist Control Group (Active Comparator): Participants will complete baseline measures 7 days prior to total knee arthroplasty and will receive a 7 week supply after completion of 12 week post-surgery visit.
  Interventions: Other: Standard Care by Surgeon and Physical Therapist

INTERVENTIONS:
Dietary Supplement: Peanut Protein Powder — Peanut protein powder will be provided to participants who will be instructed to consume 72g daily, mixed with water
  Arms: Immediate Intervention Group
Other: Standard Care by Surgeon and Physical Therapist — Patient will receive standard care from treating physicians and physical therapists pre- and post-operatively

SUMMARY:
This randomized controlled trial will study the effects of peanut protein supplementation on changes in muscle size and quality in patients undergoing total knee arthroplasty.

DETAILED DESCRIPTION:
Total knee arthroplasty (TKA) is an effective treatment for patients with knee osteoarthritis (OA) accompanied by severe pain and functional limitations. With the success of this treatment and increasing incidence of OA, it has been projected that ~3.5 million older adults will undergo TKA annually by the year 2030. While TKA is effective for reducing pain and improving health-related quality of life, TKA patients experience significant skeletal muscle atrophy and weakness in the surgical leg following surgery which, long-term, can compromise balance, functional mobility and increase fall risk. Thus, interventions to mitigate muscle atrophy and weakness post-surgery are essential to improving long-term outcomes in patients undergoing TKA.

This randomized controlled trial will study the effects of peanut protein supplementation on changes in muscle size and quality in patients undergoing total knee arthroplasty. Patients (n=30) between the ages of 60-75 years scheduled to undergo total knee arthroplasty at the Jack Hughston clinic/hospital will be recruited to participate. Participants will be stratified by gender and randomized to a peanut protein (PP) supplementation (72g daily, n=15) or waitlist control (standard care with no PP, n=15) group who will be provided with PP following the intervention. Participants in the PP group will consume PP daily starting 7 days prior to surgery and for 6 weeks post-surgery. Participants will be monitored for changes in muscle size and quality (peripheral quantitative computed tomography), upper-leg strength (isokinetic dynamometry), knee range of motion (ROM; goniometry), pain (questionnaire and pressure algometry), and functional mobility outcomes (questionnaire, timed up and go, 2-min walk test) prior to surgery and at 6 and 12-weeks post-surgery.

ELIGIBILITY:
Inclusion Criteria:

* total knee arthroplasty scheduled within two weeks under the care of surgeons at the Jack Hughston Clinic

Exclusion Criteria:

* history of invasive lower extremity surgery within the last 5 years
* allergy to peanuts or peanut products
* Body Mass Index <20 or >35 kg/m2
* currently adhering to a restrictive weight loss diet
* current or recent (within the last 2 months) steroid use
* any physical condition that interferes with performing post-surgery rehabilitation
* known peripheral vascular disease, kidney disease, liver disease, or uncontrolled endocrine disorder
* known overt cardiovascular or metabolic such as heart disease/failure or diabetes
* Radiation exposure within the last 6 months other than dental x-rays or associated with current knee treatment/diagnosis

Ages: 60 Years to 75 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult, Older Adult
Enrollment: 1 (Actual)
Dates: Start 2021-08-01 (Actual); Primary Completion 2022-04-01 (Actual); Study Completion 2022-04-01 (Actual)

PRIMARY OUTCOMES:
Change in mid-thigh skeletal muscle area | 0-6 weeks, 6-12 weeks
  peripheral quantitative computed tomography (pQCT) cross-sectional image of mid-right thigh assessed for total muscle cross-sectional area
Change in mid-thigh skeletal muscle area and quality | 0-6 weeks, 6-12 weeks
  peripheral quantitative computed tomography (pQCT) cross-sectional image of mid-right thigh assessed for overall muscle density

SECONDARY OUTCOMES:
Change in leg extensor isokinetic dynamometry | 0-6 weeks, 6-12 weeks
  maximal isokinetic right leg extensions on an isokinetic dynamometer (BioDex)
Physical Function testing | 0-6 weeks, 6-12 weeks
  3 meter up and go test
Physical Performance testing | 0-6 weeks, 6-12 weeks
  2 minute walk test
Oxford Knee Score | 0-6 weeks, 6-12 weeks
  12 question inventory
Change in inflammatory biomarkers | 0-6 weeks, 6-12 weeks
  serum C-reactive protein, interleukin-6, tumor necrosis factor-alpha, plasma 8-hydroxy-2'deoxyguanosine

CONTACTS AND LOCATIONS:
Overall Officials: Randall J Ruark, MD, Study Chair — Jack Hughston Memorial Hospital
Locations (1):
- Auburn University, Auburn, Alabama, United States

IPD SHARING:
Plan to Share IPD: No